CLINICAL TRIAL: NCT03736655
Title: Non Randomised Multi-centered Study to Evaluate Safety and Efficacy of a Novel Interposition Supraciliary Implant in Glaucoma Patients Refractory to Topical Therapy
Brief Title: Study of a Novel Interposition Supraciliary Implant in Patients With Open Angle Glaucoma
Acronym: SAFARI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Ciliatech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-FR-18-07-024848
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interposition supraciliary implant (Experimental): Any patients corresponding to inclusion / exclusion criteria
  Interventions: Device: Interposition supraciliary implant

INTERVENTIONS:
Device: Interposition supraciliary implant — Surgical placement of an interposition supraciliary implant in the supraciliary space

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a novel interposition supraciliary implant as a stand-alone therapy for lowering intraocular pressure (IOP) in patients with primary open angle glaucoma (POAG) who have failed at least one class of topical medical therapy

DETAILED DESCRIPTION:
68 patients will be included in this 5 years interventional study. All patients shall be indicated for glaucoma surgery alone (not combined with cataract), and will undergo incisional glaucoma therapy, including a novel simplified surgical technique allowing placement of an interposition supraciliary permanent device.

Several patient data like IOP, visual capacity or associated pharmacological treatments will be recorded pre and post-operatively all along the follow-up.

Purpose is to ensure device safety, and verify IOP and associated pharmacological treatment reduction after surgery, and evolution along follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POAG Schafer 3 or 4
* Medicated IOP ≥ 21

Exclusion Criteria:

* Inflammatory, congenital, traumatic, neovascular, ICE syndrome, angle closure and Schaffer 1 and 2 glaucoma
* Non surgical interventional treatment (cyclophotocoagulation, ultrasounds, …)
* Medical treatment having intraocular hypotensive effect

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Assess post-op IOP reduction | 6 months
  Proportion of Eyes With Intraocular Pressure (IOP) Reduction of ≥ 20%
Assess post-op IOP clinical success | 6 months
  Proportion of Eyes With Intraocular Pressure (IOP) < 21 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Philippe SOURDILLE, Study Director — Ciliatech
Locations (1):
- Hopital Paris Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No